CLINICAL TRIAL: NCT05581498
Title: Glaucoma Exercise as Medicine Study (GEMS).
Acronym: GEMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00336336
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLAUCOMA (Experimental): we will recruit patients with a diagnosis of primary Glaucoma for the experimental group.
  Exercise bikes and muscle-strength exercise belts will be used for exercise interventions.
  Interventions: Behavioral: Exercise, Bike exercise and muscle strength exercise.
- CONTROL (Active Comparator): we will recruit normally sighted older adults for the control group.
  Exercise bikes and muscle-strength exercise belts will be used for exercise interventions.
  Interventions: Behavioral: Exercise, Bike exercise and muscle strength exercise.

INTERVENTIONS:
Behavioral: Exercise, Bike exercise and muscle strength exercise. — Study participants will perform 12 weeks of home-based exercise training with a health bike and muscle strength exercise with a resistance belt under the supervision of a certified exercise trainer.
  The exercise will be delivered 3 days a week for 75 minutes for 12 weeks.

SUMMARY:
Project Summary Abstract:

While lifestyle changes, particularly exercise, have been suggested to protect against damage to ganglion cells in animal models, definitive evidence demonstrating its benefits in humans is lacking. Here, in a group of individuals with ganglion cell damage from glaucoma and a separate control group without significant eye disease, the investigators study the effects of a remotely delivered exercise training program by a trained exercise physiologist consisting of resistance training combined with cycling on a stationary bike. Three outcomes will be examined to evaluate if exercise might be of potential long-term benefit in protecting ganglion cells. In Aim 1, the investigators will examine the trial's primary outcome, a comparison of the pointwise change in the visual field (VF) sensitivity over the exercise period compared to a preceding usual activity period. Given the subjective nature of VF testing, Electroretinogram (ERG) testing will be employed as a more objective secondary outcome. Together, these outcomes will determine if neuro recovery is possible with exercise in individuals with GC damage from glaucoma (as has been demonstrated for Intraocular pressure (IOP)-lowering and, more recently, nicotinamide) and if neuro enhancement (improvement in the function above an already-normal level) is possible in adults without eye disease. In Aim 2, the investigators will examine if an exercise produces physiologic changes in the human eye (glaucoma and control), which would give mechanistic plausibility for a neuroprotective effect. Specifically, the investigators will compare exercise-induced changes in large vessel retinal blood flow, the density of and flux within perfused capillaries, large-vessel arterial-venous oxygen (O2) saturation gradients, inner retinal O2 metabolism, and serum levels of brain-derived neurotrophic factor (BDNF) to changes occurring in the preceding usual activity control period. Finally, in Aim 3, the investigators will examine if exercise benefits quality of life (QOL) in individuals with VF damage from glaucoma within specific domains (mobility, ocular discomfort, and mood) independent of changes in visual function. Together, these findings will provide important information regarding whether exercise produces short-term changes in eyes, which suggests possible long-term protection against ganglion cell damage.

DETAILED DESCRIPTION:
1. A. Our proposed work lies on the premise that: (1) preventing visual field (VF) damage will preserve functionality and quality of life (QoL); (2) small degrees of VF improvement are possible in eyes with ganglion cells (GC) damage (using glaucoma as a model), and therapies yielding such improvements may provide long-term neuroprotection; (3) retinal vascular parameters and neuroprotective agents (BDNF) contribute to GC damage, and therapies that improve these parameters (i.e., exercise) can prevent the onset or worsen of VF damage; and (4) QoL can be improved in patients with GC damage independent of the severity of VF damage. Based on this premise, the investigators propose to establish if exercise can create measurable improvements in GC function (Aim 1) and improve retinal vascular parameters and levels of neuroprotective factors (BDNF; Aim 2), which would suggest it may be useful in protecting against further GC damage, preserving the quality of life. Finally, the investigators also propose that exercise can improve elements of QoL independent of vision changes (Aim 3).
2. Background Several studies provided evidence that sedentary lifestyles contribute significantly to the development of a significant risk of age-related disease and complications. The investigator's previous work on 141 older adults with manifest Glaucoma and glaucoma suspects has shown slower VF loss rates with moderate-vigorous physical activity (PA) and non-sedentary activities. 2.6 hours of increased PA and additional 5000 daily steps have shown a decrease in the VF loss up to 10% in the treated group of glaucoma patients with more steps (+0.007 decibel (dB)/year/1000 daily steps, P < 0.001), moderate to vigorous activity (+0.003 decibel (dB) /year/10 more minutes of moderate-to-vigorous activity per day, P < 0.001), and more non-sedentary activity (+0.007 decibel (dB) /year/30 more minutes of non-sedentary time per day, P = 0.005). Another study demonstrated a strong association between decreased activity fragmentation with the severity of VF damage reflecting lower physiologic functions; each 5- decibel (dB) decrement in (integrated visual field) IVF sensitivity was associated with 16.3 fewer active minutes/day (P < 0.05). There is a strong need to establish the association between ocular physiology and PA; Therefore, more mechanistic approaches demonstrating the vascular physiology related to improved visual functions and neuroprotection in Glaucoma are needed. More practical methods for effective therapy and long-term randomized controlled trials are required to prove a cause-effect relationship.
3. Study design, including the sequence and timing of study procedures This study is designed as a single-center prospective study in which all subjects are evaluated over consecutive 12-week usual activity (control) and exercise (intervention) periods. This design was chosen over: (1) a cross-over design, which would be challenged by some participants assigned initially to exercise and continuing to exercise after crossing over into usual activity, or (2) a comparison of exercise and waitlist-control groups. (3) 20 normally sighted control participants aged 21 years or above will be included for pilot testing. The idea behind including the younger age group is to test the study procedure's validity and give insight into the project's true scope. Also, there is less data on how these age groups may respond to interventions being studied. The latter would require a much larger sample size (necessitating a multicenter study where the proposed imaging would not be available) due to greater across-subject vs. within-subject variability, particularly in ERG testing. Notably, ERG testing is a particularly important study outcome as it objectively measures GC function to confirm that improvements in the primary outcome measure (VF sensitivity) are not due to improved attention, cognition, or reaction speed. The investigators also include both a control (no eye disease) and glaucoma (model disease of GC damage) group, as (1) changes in GC function may occur from the recovery of damaged but alive GCs (neuro recovery) or improvement in GC function regardless of the level of damage (neuro enhancement) - a distinction that can be made only by the inclusion of normal controls; (2) improvement in physiological parameters (especially blood flow) in the control group will serve as a positive control given that improvements in retinal blood flow have been seen with a high-speed circuit resistance training program in older adults without eye disease, and (3) comparisons of exercise-related changes in the control and glaucoma groups will confirm that the putative physiological benefits of exercise are not lost in eyes with GC damage from glaucoma.

Participants will perform 6 study visits in which the participants will be evaluated by: (1) Visual fields (VFs), (2) Electroretinogram (ERG), (3) Laser speckle contrast imaging (LSCI), (4) Optical coherence tomography angiography (OCTA), (5) Visible light optical coherence tomography (VisOCT), (6) QoL using the Glaucoma computer adaptive test (GlauCAT™) and (7) fitness testing via the physical working capacity (PWC) test. Visits will occur in clustered pairs before and after the usual activity and after the exercise. During the exercise program, participants will complete three 75' exercise sessions weekly in remote groups, connected to each other and the instructor via zoom link.

The investigators will recruit 75 glaucoma patients, and 75 normally sighted controls aged 21 to 80 from the Johns Hopkins Wilmer Eye Institute to have 60 subjects in each group who pass initial entry screening and 50 in each group completing all study procedures. Glaucoma subjects will be diagnosed with primary open-angle glaucoma based on clinical exams, Optical coherence tomography (OCT) imaging, and VF testing. Evidence of glaucoma should be present in both eyes, with one eye demonstrating a mean deviation (MD) between -5 and -15 decibel (dB). Controls will be recruited from home cohabitants (spouses/partners) of patients visiting the Wilmer Eye Institute, patients seen for routine eye care (general eye exam, refraction), and, if necessary, community volunteers. Controls will be required to have normal visual acuity (VA) (20/40 or better) and contrast sensitivity (logCS>1.50) in each eye and no self-reported ocular conditions other than mild cataract, dry eye, refractive error, or other non-visually significant conditions (ocular allergies, pinguecula, etc.).

In both groups, individuals will be excluded with a history of any of the following in either eye: diabetic retinopathy, retinal detachment, uveitis, retinal artery or vein occlusion, central serous retinopathy, amblyopia, or other conditions resulting in a corrected VA worse than 20/40; controls will also be excluded if the participants have a history of glaucoma, suspect glaucoma, or ocular hypertension. Other exclusion criteria are uncontrolled blood pressure Systolic blood pressure (SBP)>160 or Diastolic blood pressure (DBP) >100), incisional surgery (ocular or non-ocular) in the past 6 months, comorbidities making exercise program impossible, cigarette smoking, body mass index (BMI) <18 or >42 kg/m2, or pregnancy. Patients reporting moderate/vigorous activity for more than 90 minutes/week will also be ineligible. Suitability for exercise will be determined using the Physical Activity Readiness Questionnaire Plus (PARQ+). Study recruitment will occur at the Johns Hopkins Wilmer Eye Institute, either the East Baltimore campus clinic, or 2 of the busiest satellite clinics - Green Spring Station and Columbia, located 12 and 24 miles from the East Baltimore campus. At least 3 of the 6 study visits will occur at the Wilmer Eye Institute East Baltimore Campus, where the Optical coherence tomography angiography (OCT-A) and visible light optical coherence tomography (Vis OCT) machines are located. The remaining study visits can be conducted at the Columbia or Green Spring Station clinics if more convenient for the patient. The exercise intervention will occur remotely over Zoom, with the exercise physiologist located in the participant's home or office and the study participant located in the participant's home.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 40 to 80 (for glaucoma and control groups - pilot subjects must be age 21-80)
2. Ability to read and respond to questions in English (facilitating GlauCAT™ questionnaire completion)
3. Physician diagnosis of primary open-angle glaucoma in both eyes (glaucoma group)
4. Visual field mean deviation between -5 and -15 dB (decibel) in at least one eye (glaucoma group)
5. Visual acuity of 20/40 or better in both eyes (control and pilot groups)
6. Normal contrast sensitivity as judged by a logCS>1.50 in both eyes (control and pilot groups)
7. Willingness to have at least 1 eye dilated at 3 prescribed study visits.

Exclusion Criteria:

1. The presence of self-reported or chart-recorded significant comorbid eye conditions in either eye, including diabetic retinopathy, retinal detachment, uveitis, retinal artery or vein occlusion, central serous retinopathy, amblyopia, or optic neuropathy other than glaucoma.
2. Individuals will also be excluded from the control group if they have a history of self-reported or chart-recorded glaucoma, suspect glaucoma, or ocular hypertension. Individuals with less serious conditions (dry eye, early cataract, mild posterior capsular opacification, mild epiretinal membranes, allergic conjunctivitis, pinguecula, etc.) will be allowed into the study if they meet the visual criteria above.
3. Uncontrolled blood pressure (BP), with systolic blood pressure (SBP) BP>160 or diastolic blood pressure (DBP) BP>100 at the first study visit (with or without anti-hypertensive medications).
4. Incisional procedures (ocular or non-ocular) in the past 6 months (minor dermatological procedures are acceptable).
5. Self-report of comorbidities or orthopedic issues which would make the prescribed exercise (resistance band training and exercise bicycling) impossible.
6. Current cigarette smoking or using electronic cigarettes to smoke.
7. Body mass index <18 or >42 kg/m2.
8. Current or planned pregnancy.
9. Self-report moderate or vigorous activity for more than 90 minutes weekly. Activities classified as moderate/vigorous include running, swimming, resistance training, most sports (basketball, volleyball, tennis), walking briskly (15' per mile), bicycling, active gardening, aerobics, or other similar activities.
10. Suitability for exercise will be confirmed by administering the Physical Activity (PA) Readiness Questionnaire Plus (PAR-Q+), a two-part questionnaire in which individuals can be categorized as fit for exercise. In the first part of the questionnaire, patients are asked 7 questions regarding self-reported: (1) heart disease/high blood pressure, (2) chest pain at rest or with activity, (3) poor balance, dizziness or loss of consciousness, (4) chronic medical conditions other than heart disease, (5) medications for chronic medical conditions, (6) bone or joint problems that could worsen with physical activity, or (7) being told by a doctor that they should only do medically-supervised physical activity.
11. If individuals answer no, they are eligible for the exercise intervention.
12. If they answer yes, they are asked several additional, more detailed questions to gauge the severity of their conditions (i.e., arthritis requiring steroid injections or tablets, cancer requiring active chemotherapy, chronic heart failure, etc.). If they answer yes to any of these questions, they will be excluded from study participation.
13. As some exclusion criteria (blood pressure, body-mass index, PAR-Q+ scores) are obtained after the consent, the numbers consenting and proceeding to the test will differ.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of VF points | Baseline, 3 months, 6 months
  Number of VF points location measurements assess the mean defect (MD) in the top quartile for rate of change during the exercise period vs. the usual activity control period as the primary outcome variables of the study.

SECONDARY OUTCOMES:
Change in ocular blood flow | Baseline, 3 months, 6 months
  The secondary outcomes will compare within-group (glaucoma, control) change in the following measures over the exercise period as compared the the usual activity period: Ocular blood flow (dynamic and static), oxygenation and vascular perfusion of the optic nerve head (ONH) and ERG PhNR.
Change in ERG photopic negative response (PhNR) | Baseline, 3 months, 6 months
  The secondary outcomes will compare within-group (glaucoma, control) change in the following measures over the exercise period as compared the the usual activity period: Ocular blood flow (dynamic and static), oxygenation and vascular perfusion of the optic nerve head (ONH) and ERG PhNR.

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Y Ramulu, MD, PHD, Principal Investigator — The Johns Hopkins University

REFERENCES:
- [Background] Lee MJ, Wang J, Friedman DS, Boland MV, De Moraes CG, Ramulu PY. Greater Physical Activity Is Associated with Slower Visual Field Loss in Glaucoma. Ophthalmology. 2019 Jul;126(7):958-964. doi: 10.1016/j.ophtha.2018.10.012. Epub 2018 Oct 10. PMID 30315900
- [Background] Stewart KJ. Physical activity and aging. Ann N Y Acad Sci. 2005 Dec;1055:193-206. doi: 10.1196/annals.1323.029. PMID 16387725
- [Background] E JY, Schrack JA, Mihailovic A, Wanigatunga AA, West SK, Friedman DS, Gitlin LN, Li T, Ramulu PY. Patterns of Daily Physical Activity across the Spectrum of Visual Field Damage in Glaucoma Patients. Ophthalmology. 2021 Jan;128(1):70-77. doi: 10.1016/j.ophtha.2020.06.053. Epub 2020 Jun 29. PMID 32615202
- [Background] Zhang J, Strand K, Totillo M, Chen Q, Signorile JF, Jiang H, Wang J. Improvement of retinal tissue perfusion after circuit resistance training in healthy older adults. Exp Gerontol. 2021 Apr;146:111210. doi: 10.1016/j.exger.2020.111210. Epub 2020 Dec 29. PMID 33385483
- [Background] Cardinal BJ, Esters J, Cardinal MK. Evaluation of the revised physical activity readiness questionnaire in older adults. Med Sci Sports Exerc. 1996 Apr;28(4):468-72. doi: 10.1097/00005768-199604000-00011. PMID 8778552